CLINICAL TRIAL: NCT02127580
Title: Balloon Expandable Transcatheter Aortic Valve Implantation Without Predilation of the Aortic Valve (EASE-IT) A Two-armed Registry
Brief Title: Balloon Expandable Transcatheter Aortic Valve Implantation Without Predilation of the Aortic Valve
Acronym: EASE-IT
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: EASE-IT
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Aortic Valve Stenosis
Keywords: THV; BAV; pre-dilation; Aortic valve stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with BAV: Patients undergoing TA-TAVI WITH predilation of the AV (Group A)
  Interventions: Procedure: BAV
- without BAV: Patients undergoing TA-TAVI WITHOUT predilation of the AV
  Interventions: Procedure: without BAV

INTERVENTIONS:
Procedure: BAV
  Groups: with BAV
Procedure: without BAV
  Groups: without BAV

SUMMARY:
There is limited experience for the balloon expandable THV (transcatheter heart valve) on the need for predilation (ballon aortic valvuloplasty, BAV). Therefore we aim to verify results of a small case series published by Wendler et. al. to examine hard endpoints such as the incidence of cerebrovascular complications, paravalvular leakage and operative outcomes in a multicenter registry.

We aim to compare the implantation of balloon expandable transcatheter heart valves with or without predilation with respect to procedural outcomes (VARC2).

DETAILED DESCRIPTION:
Prior to the deployment of transcatheter heart valves (THV), balloon aortic valvuloplasty (BAV) is usually performed under rapid right ventricular pacing (burst >180 bpm) with the induction of a functional cardiac arrest for up to 30 seconds. Aortic valve predilation is aiming at facilitating the crossing of the aortic annulus, accurate valve positioning and does also provide information on the anatomy of the valve complex. However, BAV has been shown to have a number of potentially detrimental effects, such as:

* Functional cardiac arrest induced by rapid pacing leads to transient coronary, cerebral, and renal ischemia.
* In patients with a reduced left ventricular ejection fraction (LVEF), prolonged cardiac depression after rapid pacing is observed and may result in hemodynamic failure and systemic inflammatory response syndrome (SIRS). Both are associated with a high periprocedural mortality.
* BAV has been identified as a major source of thrombotic and valvular material and increases the risk for coronary obstruction with subsequent myocardial infarction and stroke.
* The local trauma in the left-ventricular outflow tract caused by BAV may potentially contribute to aortic root rupture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for TAVI as to the Edwards THV IFU
* Eligible for TABI with AND without BAV
* Signed informed consent

Exclusion Criteria:

* Logistic EuroSCORE I >50%
* Mitral or tricuspid valvular insufficiency (> grade II)
* Previous aortic valve replacement
* Uncontrolled atrial fibrillation
* Left ventricular or atrial thrombus by echocardiography
* Recent cerebrovascular event (within the last 3 months)
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from aortic Stenosis undergoing transapical trans-catheter heart valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
VARC2 criteria | 3 months
  comparison of the implantation of balloon expandable transcatheter heart valves with or without predilation with respect to procedural outcomes (VARC2).

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schröfel, MD, Principal Investigator — Clinic for Cardiac Surgery Karlsruhe; Justus Strauch, Prof., Principal Investigator — Klinik für Herz- und Thoraxchirurgie
Locations (7):
- Germany (7):
  - Clinic for Cardiac Surgery Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Klinik für Herz- und Thoraxchirurgie, BG-Uniklinikum Bergmannsheil, Bochum, North Rhine-Westphalia
  - Klinikum Augsburg, Augsburg
  - Herz- und Gefäß-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale
  - Schüchtermann-Schiller'sche Kliniken, Bad Rothenfelde
  - Uniklinik Köln, Cologne
  - Uniklinik Essen, Essen

REFERENCES:
- [Result] Strauch J, Wendt D, Diegeler A, Heimeshoff M, Hofmann S, Holzhey D, Oertel F, Wahlers T, Kurucova J, Thoenes M, Deutsch C, Bramlage P, Schrofel H. Balloon-expandable transapical transcatheter aortic valve implantation with or without predilation of the aortic valve: results of a multicentre registry. Eur J Cardiothorac Surg. 2018 Apr 1;53(4):771-777. doi: 10.1093/ejcts/ezx397. PMID 29182764
- [Derived] Bramlage P, Strauch J, Schrofel H. Balloon expandable transcatheter aortic valve implantation with or without pre-dilation of the aortic valve - rationale and design of a multicenter registry (EASE-IT). BMC Cardiovasc Disord. 2014 Nov 18;14:160. doi: 10.1186/1471-2261-14-160. PMID 25403092